CLINICAL TRIAL: NCT00599508
Title: Nutritional Supplementation in Cognitive Aging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Welch Foods Incorporated (Industry); U.S. Highbush Blueberry Council (Other)
Responsible Party: Principal Investigator, Robert Krikorian, Clinical Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 06-03-20-08
Record Dates: First submitted 2008-01-10; First posted 2008-01-23 (Estimated); Last update posted 2016-10-10 (Estimated); Status verified 2016-10

CONDITIONS: Cognitive Aging
Keywords: memory; aging

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- grape juice active intervention (Active Comparator): Concord grape juice administered daily for 12 or 16 weeks
  Interventions: Dietary Supplement: Concord grape juice
- juice placebo (Placebo Comparator): berry placebo juice administered daily for 12 or 16 weeks
  Interventions: Dietary Supplement: placebo juice
- blueberry juice active intervention (Active Comparator): wild blueberry juice administered daily for 12 weeks
  Interventions: Dietary Supplement: blueberry juice
- blueberry powder intervention (Active Comparator): whole fruit blueberry powder administered daily for 16 weeks
  Interventions: Dietary Supplement: whole fruit blueberry powder
- powder placebo (Placebo Comparator): placebo powder administered daily for 16 weeks
  Interventions: Dietary Supplement: berry placebo powder

INTERVENTIONS:
Dietary Supplement: Concord grape juice — Several ounces Concord grape juice administered 3 times a day for 12 or 16 weeks. Specific dosage determined by participant's weight.
  Other Names: Welch's Concord Grape Juice
  Arms: grape juice active intervention
Dietary Supplement: placebo juice — several ounces placebo juice consumed three times a day for 12 or 16 weeks; dosage determined according to participant's weight
  Arms: juice placebo
Dietary Supplement: blueberry juice — wild blueberry juice administered daily for 12 weeks, dosage determined according to participant's weight
  Arms: blueberry juice active intervention
Dietary Supplement: whole fruit blueberry powder — whole fruit, freeze dried blueberry powder derived from a blend of cultivated blueberries administered daily for 16 weeks
  Arms: blueberry powder intervention
Dietary Supplement: berry placebo powder — berry placebo powder administered daily for 16 weeks
  Arms: powder placebo

SUMMARY:
To evaluate the effect of supplemented berry fruit juice and whole fruit berry powder on memory performance and brain function in older adults

DETAILED DESCRIPTION:
Randomized trials involving daily supplementation with berry fruits in older adults with early memory changes. The berry products include Concord grape juice, blueberry juice, and whole fruit blueberry powder. Supplementation periods are 12 and 16 weeks, depending on berry product. The Aims of the studies are to assess effects on cognitive performance and in a subset of participants, in brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Mild Cognitive Impairment

Exclusion Criteria:

* Diabetes
* Weight of under 100 or over 210 pounds
* Chronic use of pain medication

Min Age: 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2006-06; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
memory performance | at the end of the intervention

SECONDARY OUTCOMES:
cortisol | at the end of the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Robert Krikorian, Ph.D., Principal Investigator — University of Cincinnati
Locations (1):
- University of Cincinnati, Cincinnati, Ohio, United States